CLINICAL TRIAL: NCT04058821
Title: Novel MRI for Diagnosing Traumatic Brachial Plexus Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PL18/110632
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with traumatic brachial plexus injuries (Experimental): Participants will have two MRI scans before surgery (to find out the best time to scan), then two after surgery (at 6 and 12 months).
  Interventions: Diagnostic Test: Novel MRI scan - 7 days post injury; Diagnostic Test: Novel MRI scan - 14 days post injury; Diagnostic Test: Functional MRI scan - 6 months post brachial plexus exploration; Diagnostic Test: Functional MRI scan - 12 months post brachial plexus exploration

INTERVENTIONS:
Diagnostic Test: Novel MRI scan - 7 days post injury — * A turbo spin-echo localiser (20 seconds)
  * Single-shot echo planar diffusion tensor imaging (7 minutes)
  * 3D constructive interference in steady state (CISS, 6 minutes)
  * Phase-sensitive inversion-recovery gradient echo with cardiac gating (4 minutes)
Diagnostic Test: Novel MRI scan - 14 days post injury — * A turbo spin-echo localiser (20 seconds)
  * Single-shot echo planar diffusion tensor imaging (7 minutes)
  * 3D constructive interference in steady state (CISS, 6 minutes)
  * Phase-sensitive inversion-recovery gradient echo with cardiac gating (4 minutes)
Diagnostic Test: Functional MRI scan - 6 months post brachial plexus exploration — * Continuous whole brain echo-planar imaging
  * High-resolution T1-weighted imaging of the brain
  * Bilateral magnetic resonance spectroscopy (12 minutes)
Diagnostic Test: Functional MRI scan - 12 months post brachial plexus exploration — * Continuous whole brain echo-planar imaging
  * High-resolution T1-weighted imaging of the brain
  * Bilateral magnetic resonance spectroscopy (12 minutes)

SUMMARY:
The aims are:

1. Investigate new magnetic resonance imaging (MRI) scans for diagnosing severe nerve injury in the arm.
2. Understand how the brain and spinal cord respond to severe nerve injury using MRI.

The nerves which control movement and feeling in the arm can be severely damaged in eg. motorbike crashes, sporting or work-related injuries. Every year 500 adults sustain life-changing major nerve injuries, causing 1) disability needing constant care, 2) life-long pain and 3) mental illness. In England, major nerve injuries cost £250million every year in hospital treatments, unemployment and social care. Injured nerves can be repaired with surgery.

To decide if nerves need repairing, exploratory surgery is needed. Instead, we have developed a new MRI scan which could diagnose nerve injuries, meaning that exploratory surgery could be avoided, nerve injuries could be diagnosed sooner and reconstructive surgery performed sooner.

Some people with nerve injuries develop lifelong pain - if we could understand how the brain adapts, we could learn how to prevent nerve pain. Also, some people don't recover movement in their hand - if we could understand how the brain reorganises nerves controlling movement, we could predict who would benefit from surgery.

ELIGIBILITY:
Inclusion Criteria:

Adults with traumatic BPIs who require surgical exploration of the supraclavicular brachial plexus. A traumatic BPI is defined by the absence of any or all motor or sensory function in an upper limb, following trauma.

Exclusion Criteria:

* Patients with an acutely ischaemic limb as they require immediate surgical intervention
* Unable to get into the MRI scanner due to habitus or claustrophobia
* Unable to lie still due to any cause (eg. athetoid movements, dystonias, chorea, etc)
* Intraocular or intracranial metallic foreign bodies
* Active implants (eg. pacemakers, implantable cardiac defibrillators, nerve stimulators, etc) which are not MRI safe or conditional.
* Pregnancy - whilst there are no known adverse effects of MRI(129-131) to the mother or fetus, MRI is generally avoided in pregnancy due to the acoustic trauma(132) and inductive heating generated by alternating magnetic fields.
* Any pre-existing neurological disorder, injury or disease causing a functional impairment in the affected limb
* Patients lacking capacity to consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of diffusion tensor MRI for detecting any root avulsion of the brachial plexus | 7 mins
  diagnostic accuracy of diffusion tensor MRI for detecting any root avulsion of the brachial plexus

CONTACTS AND LOCATIONS:
Locations (1):
- St James's University Hospitals NHS Trust, Leeds, United Kingdom